CLINICAL TRIAL: NCT05976633
Title: Evaluating the Factors That Influence Glycemic Response to Wild Rice and Wild Rice Blends in Humans (EFGW) Study.
Brief Title: Glycemic Response to Wild Rice and Wild Rice Blends in Humans Study
Acronym: EFGW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HS25900 (B2023:033)
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Blood Glucose
Keywords: glycemic response; glycemic control; rice

STUDY DESIGN:
Intervention Model Description: crossover randomized clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Consumption of 1 of 3 rice products (Experimental): This arm will provide 1 of the 3 randomly assigned rice products to the participant and there will be a minimum of three days separating each visit.
  Interventions: Other: 15% Wild rice and 85% Brown rice blend - Stovetop
- Consumption of 2 of 3 rice products (Experimental): This arm will provide the consumption of the second randomly assigned rice product. There will be a minimum of three days separating each visit.
  Interventions: Other: Whole wild rice
- Consumption of 3 of 3 rice products (Experimental): This arm will provide the third consumption of the randomly assigned rice product. There will be a minimum of three days separating each visit.
  Interventions: Other: Whole brown rice
- Consumption of the control rice product (Active Comparator): This arm will provide the white rice control product.
  Interventions: Other: Whole white rice (control)
- Consumption of 1 of 3 rice products with different preparation method (Experimental): This arm will provide the blends product via a different cooking method (microwave).
  Interventions: Other: 15% Wild rice and 85% Brown rice blend - Microwaved

INTERVENTIONS:
Other: Whole white rice (control) — One serving size (140g cooked on stovetop) of whole white rice will be provided. Cooking time will be consistently maintained throughout.
  Arms: Consumption of the control rice product
Other: Whole brown rice — One serving size (140g cooked on stovetop) of whole brown rice will be provided. Cooking time will be consistently maintained throughout.
  Arms: Consumption of 3 of 3 rice products
Other: Whole wild rice — One serving size (140g cooked on stovetop) of whole wild rice will be provided. Cooking time will be consistently maintained throughout.
  Arms: Consumption of 2 of 3 rice products
Other: 15% Wild rice and 85% Brown rice blend - Stovetop — One serving size (140g cooked on stovetop) of 15% wild rice and 85% brown rice blend (Myera) will be provided. Cooking time will be consistently maintained throughout.
  Arms: Consumption of 1 of 3 rice products
Other: 15% Wild rice and 85% Brown rice blend - Microwaved — One serving size (140g cooked in microwave) of 15% wild rice and 85% brown rice blend (Myera) will be provided. Cooking time will be consistently maintained throughout.
  Arms: Consumption of 1 of 3 rice products with different preparation method

SUMMARY:
The goal of this clinical trial is to test the effects of wild rice and wild rice blends compared to other rice on glycemic control and evaluating factors that influence glycemic response to wild rice in healthy individuals. The main questions aim to answer:

1. Is there an effect of wild rice on blends on glycemic control and response?
2. Does cooking wild rice via stovetop or microwave change its glycemic response?
3. Is the wild rice blend product palatable?
4. What is the subjective appetite when consuming the treatment?

Participants will:

* consent to attend 5 study visits being 2.5 hours each
* come to each visit fasted for at least 10-12 hours.
* complete a Motivation to Eat VAS following each blood measure

DETAILED DESCRIPTION:
This study will be a crossover randomized trial consisting of 5 sessions. The wild rice products will be provided by the Myera group.

Participants will fast and arrive at the Richardson Centre for Food Technology and Research (RCFTR) between 7am - 11am on the session day. They will be provided either of the study treatments based on randomization sequence. Baseline blood glucose (0 min) will be measured twice via finger stick blood sample right before their first bite of the study product, and at 15, 30, 45, 60, 90 and 120 mins after baseline in duplicate. VAS will be completed following consumption of the treatments to measure palatability and subjective appetite at baseline (0 min), and at 15, 30, 45, 60, 90, and 120 minute time points.

The primary objective is to test the effects of wild rice and wild rice blends compared to other rice on glycemic control and evaluating factors that influence glycemic response to wild rice in humans performed via the finger stick blood glucose that will be measured throughout each session as outlined above. Secondly, to test whether wild rice glycemic response is affected based on cooking method.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female between 18-50 years old
* BMI range in between 18.9-29.9 kg/m2
* Fasting glucose <5.6 mmol/L
* Usually eat breakfast
* Participant must receive at least two doses of COVID-19 vaccine that have been recognized by Winnipeg Regional Health Authorities.
* In the Investigator's opinion is able and willing to comply with all trial requirements

Exclusion Criteria:

* Fasting glucose ≥ 5.6 mmol/L or <3.5 mmol/L
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Participants who indicate that they could not finish study treatments within 10 minutes
* Use of medication or supplements that may influence carbohydrate metabolism, including, not limit to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of screening visit
* History of disordered eating, AIDS, hepatitis, a history of clinically important endocrine (including Type I and Type II diabetes mellitus), cardiovascular (including but not limit to atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders
* Intolerance or allergic reaction to rice
* Existing restrictive dietary habits (such a vegan, low carbohydrate/keto)
* History of hypertension
* History of cancer within the last two years (except for non-melanoma skin cancer)
* Recent history (within 12 month of screening) or current consumption of >14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Body weight change over 3.5kg for the past 3 months
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Had significant physical trauma or major surgery in the past 3 month or had trauma or major surgery in the past 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Glycemic response | Capillary blood glucose will be measured at 0 (baseline) and then 15, 30, 45, 60, 90 and 120 minutes after the treatment has been consumed..
  Finger stick blood glucose will be taken throughout each session.

SECONDARY OUTCOMES:
Palatability of rice products | VAS measurements at 0 (baseline) and then 15, 30, 45, 60, 90 and 120 minutes
  Visual Analogue Scale (VAS) assessment following consumption of the treatment
Subjective appetite | VAS measurements at 0 (baseline) and then 15, 30, 45, 60, 90 and 120 minutes.
  Visual Analogue Scale (VAS) assessment following consumption of the treatment measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan MacKay, PHD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Center for Food Technology and Research, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No